CLINICAL TRIAL: NCT03827148
Title: Impact of Pharmacist Intervention on Disease Knowledge, Rehabilitation and Medication Adherence, Treatment Induced Direct Cost, Health-related Quality of Life and Satisfaction in Patients With Rheumatoid Arthritis: a Randomized Single-blind Two-arm Controlled Trial
Brief Title: Impact of Pharmacist Intervention on Disease Knowledge, Rehabilitation and Medication Adherence, Treatment Induced Direct Cost, Health-related Quality of Life and Satisfaction in Patients With Rheumatoid Arthritis
Acronym: DRAMATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Clifton Central Hospital (Unknown)
Responsible Party: Principal Investigator, Atta Abbas Naqvi, Dr Atta Abbas Naqvi, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: USM
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Pharmacist intervention; Disease knowledge; Medication adherence; Rehabilitation; Physical therapy; Health related quality of life; Direct cost of treatment; Rheumatoid arthritis; Pakistan; Out-patients
MeSH Terms: conditions — Arthritis, Rheumatoid; Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: This study is a randomized single-blind parallel trial. The patients who participate in this study after signing of consent would be randomly assigned to either control group (CG), i.e., usual care or intervention group (IG), i.e., pharmaceutical care. The allocation ratio will be 1:1. The participants in the intervention group would be counselled by pharmacist, provided a disease education literature and would have access to pharmacist for 90 days via telephone. The participants in the control group would received usual care without pharmacist intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators, data collectors, study observers, data entry operators and data analysis statistician will be blinded to the allocation. The patients in the control group will be blinded to pharmacists as they would not know if the person they find in the room is a pharmacist or, a data collector. Similarly, the data collector would not know if the patient belong to IG or CG. However, the patients enrolled in intervention group will not be blinded to the pharmacist considering the nature of intervention yet, the pharmacist will be blinded to the outcome assessment so that there will be less likelihood of intervention bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Pharmacist-delivered pharmaceutical care (Experimental): The intervention consist of a pharmacist providing pharmaceutical care with aim to improve the treatment outcomes. It will be in the form of a single face-to-face session by pharmacist. Moreover, a specially designed rheumatoid arthritis disease education literature will be provided in both Urdu and English languages to patients for home use. The patients will be provided a contact number at which the pharmacist will be available at all times for the next three months (week 12). A specially designated counselling area in the pharmacy department of the hospitals served as venues for intervention.
  Interventions: Other: Pharmaceutical Care
- Control: Usual Care (No Intervention): The patient in control group will have usual care without pharmacist intervention.

INTERVENTIONS:
Other: Pharmaceutical Care — Pharmaceutical care is an individualized patient-centric health service delivered by pharmacists that incorporates, but is not limited to, disease education, therapy management, self-care and self-management of disease and therapy as well as motivational guidance.
  Arms: Intervention: Pharmacist-delivered pharmaceutical care

SUMMARY:
The objective of this study was to evaluate effectiveness of pharmacist intervention in improving disease knowledge, adherence to treatment, health related quality of life and direct cost of treatment. The study also documented patient satisfaction with pharmacist counselling as a quality control measure.

This is a randomized controlled single-blind two-arm trial in patients with rheumatoid arthritis in Karachi, Pakistan. The study will enroll patients with established diagnosis of rheumatoid arthritis over three months. The patients after signing written consent would be randomized through a computer-generated list in control group, i.e., usual care and intervention group, i.e., pharmaceutical care with a ratio of 1:1. The study will take place in three patient-visits over the course of three months. The patients would be intervened by pharmacist in intervention group while those in control group will have usual care. Primary outcomes include change in mean score at follow-up, i.e., week 12, for disease knowledge, adherence to medications and rehabilitation/physical therapy, health related quality of life (HRQoL). The secondary outcomes include change in the mean direct cost of treatment and patient satisfaction from pharmacist counselling.

This is a novel study that evaluates the role of pharmacist in improving treatment outcomes of patients with rheumatoid arthritis. The results of this trial could set the foundation for future delivery of care for such patients in Pakistan. The results of this trial would be published in a peer-reviewed journal.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic inflammatory disease that mainly affects the joints and results in pain, swelling and decreased mobility. The disease over the course of time, leads to joint deformity and disability. The disease ranks third as major cause of disability after osteoarthritis and gout and affects roughly 1% of global population. Decrease mobility in patients results in decreased productivity and further worsens their quality of life. While pharmacological treatment may be essential in managing the acute flares and episodic pain associated with the disease, self-care and home-based management of RA is another important area of care which patients need to incorporate to manage it effectively.

Several studies have reported that self-care in RA effectively reduces acute flares. This could be done through the use of patient education and counselling. Pharmacist provide pharmaceutical care that incorporates these areas of care. Pharmaceutical care is an individualized patient-centric health service delivered by pharmacists that incorporates, but is not limited to, disease education, therapy management, self-care and self-management of disease and therapy as well as motivational guidance.

Evidence from several randomized trials indicate that patient counselling, disease education and telephonic interventions have improved self-care practices of patients. Educating patients about managing RA empowers them in understanding signs and symptoms of disease and devise ways to reduce or limit aggravating factors. A randomized trial conducted by Petkova that involved community pharmacy-based patient education program improved treatment outcomes of arthritis patients. Moreover, Mary and colleagues demonstrated positive effect of mobile phone short message service on medication adherence of patients with RA.

In the last decade there has been only few studies that have evaluated the impact of pharmacist-led pharmaceutical care on treatment outcomes in patients with rheumatoid arthritis. In Pakistan, no study has been conducted till date that evaluates the same. Since, the disease prevalence has increased in Pakistani population of late, and mainly affects the middle-aged individuals, it is expected to affect their productivity, employ-ability and income. This would worsen their health-related quality of life and adds to economic burden of this disease on the society. Therefore, a need was felt to evaluate the impact of pharmacist-delivered pharmaceutical care on treatment outcomes in Pakistani patients with rheumatoid arthritis.

ELIGIBILITY:
Types of participants Inclusion criteria

The patients who meet the following criteria would be invited to participate in our study:

1. Patients suffering from rheumatoid arthritis diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR criteria.
2. Patients diagnosed with RA based on above mentioned criteria for at least 3 months prior to invitation.
3. Patients aged above 18 years
4. Patients visiting out-patient clinics only. Before enrolling in the study, patients attended a study explanation session and provided a written consent to participate.

Exclusion criteria

Patients were excluded from the study if they had any of the following conditions:

1. Patients with musculoskeletal illnesses other than rheumatoid arthritis
2. Patients with a recent history of surgery or planned surgery for rheumatoid arthritis
3. Patients with more than three co-morbidities
4. Patients with any lab abnormalities, being treated for liver or kidney disease
5. Patients who have had a severe infection and have completed antibiotic course in the last week
6. Patients with advanced cardiovascular disease, severe allergies or a rare disease
7. Patients who are currently participating in other clinical trial or have participated in the last three months.
8. Pregnant patients, planning to become pregnant, breast feeding and females with other gynecological issues were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Rheumatoid arthritis disease knowledge | 3 months
  Patient knowledge regarding rheumatoid arthritis will be assessed after three months (week 12) from baseline (week 0). The Rheumatoid Knowledge Assessment Scale (RAKAS) will be used to measure rheumatoid arthritis disease knowledge. The RAKAS is a thirteen-item scale that contains questions related to knowledge, symptoms, treatment and risk factors. The items are multiple choice questions (MCQs) and correct answer awards a score while the wrong answers provides no score. A cumulative score is calculated which is interpreted as excellent, good, low and poor knowledge.
Treatment adherence | 3 months
  Patient adherence to rehabilitation/physical therapy after three months (week 12) from baseline (week 0). The assessment of adherence to rehabilitation/physical therapy, will be done through Urdu version of General Rehabilitation Adherence Scale (GRAS).
Medication adherence | 3 months
  Patient adherence to medication therapy after three months (week 12) from baseline (week 0). For the assessment of adherence to medication and pharmacotherapy, the Urdu version of General Medication Adherence Scale (GMAS) will be used.
Health related quality of life (HRQoL) | 3 months
  It will be assessed after three months (week 12) from baseline (week 0).The EQ-5D-5L is a generic tool to measure health and provides a numeric value for health status of patient. The score is then calculated as per the criteria specified by the EuroQol.

SECONDARY OUTCOMES:
Direct cost of treatment | 3 months
  The mean direct cost of rheumatoid arthritis treatment after three months (week 12) from baseline (week 0) in patients enrolled in control (CG) and intervention groups (IG).
Patient satisfaction | 3 months
  Patient satisfaction resulting from pharmacist-led pharmaceutical care. The proportion (%) of patients in the intervention group (IG) who were satisfied with the intervention after three months (week 12) from baseline (week 0).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hassali, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- Clifton Central Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naqvi AA, Hassali MA, Naqvi SBS, Aftab MT. Impact of pharmacist educational intervention on disease knowledge, rehabilitation and medication adherence, treatment-induced direct cost, health-related quality of life and satisfaction in patients with rheumatoid arthritis: study protocol for a randomized controlled trial. Trials. 2019 Aug 9;20(1):488. doi: 10.1186/s13063-019-3540-z. PMID 31399128